CLINICAL TRIAL: NCT07116863
Title: A Randomized, Double-Blind, Multi-Center, Phase III Trial to Evaluate the Efficacy and Safety of KDF1901 in Patients With Essential Hypertension Inappropriately Controlled on KDF1901-R0 Treatment
Brief Title: A Multicenter, Randomized, Double-Blind Phase 3 Trial of KDF1901 in Patients With Essential Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyungdong Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KDF1901-3H
Record Dates: First submitted 2025-08-07; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KDF1901 group (Experimental): Run-in Period (4 weeks): KDF1901-R0, a fixed-dose combination tablet containing valsartan 80 mg and amlodipine 5 mg, administered once daily
  Treatment Period 1 (2 weeks): KDF1901-L, containing valsartan 80 mg, amlodipine 5 mg, and chlorthalidone 12.5 mg, administered once daily
  Treatment Period 2 (6 weeks): KDF1901, containing valsartan 160 mg, amlodipine 10 mg, and chlorthalidone 25 mg, administered once daily
  Interventions: Drug: KDF1901-R0; Drug: KDF1901-L; Drug: KDF1901
- Dual Therapy group (Active Comparator): Run-in Period (4 weeks): KDF1901-R0, a fixed-dose combination tablet containing valsartan 80 mg and amlodipine 5 mg, administered once daily
  Treatment Period 1 (2 weeks): KDF1901-R0, same as above, administered once daily
  Treatment Period 2 (6 weeks): KDF1901-R1, containing valsartan 160 mg and amlodipine 10 mg, administered once daily
  Interventions: Drug: KDF1901-R0; Drug: KDF1901-R1

INTERVENTIONS:
Drug: KDF1901-R0 — Fixed-dose combination tablet containing valsartan 80 mg and amlodipine 5 mg. Orally administered once daily for 4 weeks during the run-in period, and for 2 weeks during Treatment Period 1(Dual Therapy group).
Drug: KDF1901-L — Fixed-dose combination tablet containing valsartan 80 mg, amlodipine 5 mg, and chlorthalidone 12.5 mg.
  Orally administered once daily for 2 weeks during Treatment Period 1.
  Arms: KDF1901 group
Drug: KDF1901 — Fixed-dose combination tablet containing valsartan 160 mg, amlodipine 10 mg, and chlorthalidone 25 mg.
  Orally administered once daily for 6 weeks during Treatment Period 2.
  Arms: KDF1901 group
Drug: KDF1901-R1 — Fixed-dose combination tablet containing valsartan 160 mg and amlodipine 10 mg. Orally administered once daily for 6 weeks during Treatment Period 2.
  Arms: Dual Therapy group

SUMMARY:
This randomized, double-blind, multicenter phase 3 clinical trial evaluated the efficacy and safety of KDF1901, a single-pill triple combination of valsartan, amlodipine, and chlorthalidone, in patients with essential hypertension inadequately controlled with dual therapy. A total of 286 patients who remained uncontrolled after a 4-week run-in period with valsartan/amlodipine were randomized to receive either KDF1901 (valsartan/amlodipine/chlorthalidone 160/10/25 mg) or a dual combination of valsartan/amlodipine (160/10 mg) for 8 weeks.

The primary endpoint was the change in mean sitting systolic blood pressure (MSSBP) from baseline at week 8. Secondary outcomes included changes in diastolic BP (MSDBP), blood pressure normalization rate, and response rate. KDF1901 demonstrated significantly greater reductions in both MSSBP and MSDBP, with higher normalization and response rates compared to dual therapy. The treatment was well tolerated, and the incidence of adverse events was comparable between groups.

DETAILED DESCRIPTION:
Achieving optimal blood pressure control remains a clinical challenge, especially in patients who do not respond adequately to dual antihypertensive therapy. This study assessed the clinical benefit of adding chlorthalidone to a fixed-dose combination of valsartan and amlodipine to form KDF1901, a triple combination therapy.

The study included 286 patients with essential hypertension who did not reach target blood pressure after a 4-week run-in period with valsartan/amlodipine (80/5 mg). They were randomized 1:1 to receive either KDF1901 (160/10/25 mg) or valsartan/amlodipine (160/10 mg) for 8 weeks.

At week 8, the KDF1901 group showed significantly greater reductions in MSSBP (-21.2 ± 9.3 mmHg vs. -15.4 ± 8.7 mmHg, p<0.001) and MSDBP (-12.2 ± 6.5 mmHg vs. -8.6 ± 6.2 mmHg, p<0.001) than the dual therapy group. Blood pressure normalization and response rates were also significantly higher with KDF1901.

Subgroup analyses revealed consistent efficacy in elderly and diabetic patients. The incidence of TEAEs was similar between groups, and most adverse events were mild and not drug-related. These results suggest the potential clinical utility of chlorthalidone-based triple therapy in high-risk hypertensive patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants aged ≥19 years at the time of screening.
2. Participants who meet one of the following blood pressure criteria at screening:

   1. If not currently receiving antihypertensive medication for at least 4 weeks (treatment-naïve):

      * Mean Sitting Systolic Blood Pressure (MSSBP) ≥160 mmHg and <200 mmHg
   2. If currently receiving antihypertensive medication:

      * MSSBP ≥140 mmHg and <200 mmHg
      * For participants with cardiovascular disease, diabetes mellitus, or microalbuminuria (e.g., persistent proteinuria or hematuria), the range is:

   MSSBP ≥130 mmHg and <200 mmHg
3. Willing and able to provide written informed consent prior to participation in the study.
4. At baseline (Visit 3), participants must have MSSBP ≥140 mmHg and <200 mmHg.

   * For participants with cardiovascular disease, diabetes mellitus, or microalbuminuria: MSSBP ≥130 mmHg and <200 mmHg
5. At least 70% compliance with run-in period medication, as assessed by tablet count.

Exclusion Criteria:

1. Mean sitting diastolic blood pressure (MSDBP) ≥110 mmHg at screening (Visit 1) or baseline (Visit 3)
2. Difference in blood pressure between arms: MSSBP ≥20 mmHg and MSDBP ≥10 mmHg at screening
3. History or presence of secondary hypertension or suspected secondary hypertension, including:

   * Aortic coarctation, pheochromocytoma, Cushing's syndrome, hyperaldosteronism, polycystic kidney disease
4. Severe pulmonary, cardiac, or vascular conditions, such as:

   * Pulmonary hypertension, severe heart failure (NYHA class III or IV), hypertrophic cardiomyopathy, aortic aneurysm, thrombocytopathy
5. History of serious cardiovascular events or interventions within 24 weeks prior to screening:

   * Myocardial infarction, unstable angina, coronary revascularization (PCI/CABG)
6. History of cerebrovascular disorders within 24 weeks prior to screening:

   * Stroke, TIA, cerebral hemorrhage
7. History of ocular conditions within 24 weeks prior to screening:

   * Retinal hemorrhage, optic neuropathy, severe visual impairment
8. History of malignancy within 5 years prior to screening, except:

   * Successfully treated and in remission for ≥2 years, or
   * Basal cell carcinoma or squamous cell carcinoma of the skin
9. Hereditary blood disorders or history of angioedema related to ACE inhibitors or ARBs
10. History of galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption
11. Diagnosis of inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis) within 48 weeks prior to screening
12. Clinically significant conditions affecting drug absorption, distribution, metabolism, or excretion
13. Symptoms of orthostatic hypotension or risk of falls or syncope
14. Severe anemia, leukopenia, or thrombocytopenia at screening
15. Heart failure NYHA class III or IV
16. Known serious arrhythmias, including ventricular tachycardia or fibrillation
17. Known autoimmune disease or connective tissue disorder
18. Clinically significant renal, hepatic, or cardiovascular disease
19. eGFR <30 mL/min/1.73 m² or serum creatinine ≥2.0 mg/dL
20. ALT or AST >3× upper limit of normal (ULN)
21. Serum K+ <3.5 or >5.5 mmol/L, Na+ <135 mmol/L, Ca2+ >10.5 or <2.63 mmol/L
22. Requiring long-term immunosuppressive therapy or systemic corticosteroids
23. Clinically significant chronic inflammatory conditions
24. History of major surgery or active GI disorders
25. Type 2 diabetes mellitus with HbA1c ≥9.0%
26. Known edematous disorders (e.g., untreated nephrotic syndrome)
27. Requirement for prohibited medications (emergency drugs) during study period (Visit 1-6)
28. Use of lithium therapy
29. Use of terfenadine or astemizole
30. Hypersensitivity to study drugs, dihydropyridine-class CCBs, thiazide diuretics, or sulfonamides
31. History or suspicion of drug or alcohol abuse
32. Pregnancy or lactation
33. Women of childbearing potential or male participants not agreeing to use reliable contraception during study
34. Participation in other clinical trials or use of investigational products within 4 weeks prior to screening
35. Judged by the investigator to be otherwise unsuitable for study participation

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Actual)
Dates: Start 2022-06-21 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-09-13 (Actual)

PRIMARY OUTCOMES:
Change in Mean Sitting Systolic Blood Pressure (MSSBP) from baseline to Week 8 | Baseline to Week 8
  Mean change in sitting systolic blood pressure (MSSBP) after 8 weeks of treatment, measured at trough using a validated automated device.

SECONDARY OUTCOMES:
Change in Mean Sitting Systolic Blood Pressure (MSSBP) from baseline to Week 8 | Baseline to Week 2 and Week 4
  Mean change in MSSBP after 2 and 4 weeks of treatment, compared to baseline.
Change in Mean Sitting Diastolic Blood Pressure (MSDBP) from baseline to Week 2, Week 4, and Week 8 | Baseline to Week 2, Week 4, and Week 8
  Mean change in MSDBP measured at trough using an automated device.
Proportion of subjects achieving target blood pressure at Weeks 2, 4, and 8 | Week 2, Week 4, and Week 8
  Proportion of subjects achieving MSSBP <140 mmHg and MSDBP <90 mmHg. For subjects with diabetes mellitus, target BP is MSSBP <130 mmHg and MSDBP <80 mmHg.
Response rate at Weeks 2, 4, and 8 | Week 2, Week 4, and Week
  Proportion of subjects who achieved a reduction of ≥20 mmHg in MSSBP or ≥10 mmHg in MSDBP from baseline.

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - CHA Gangnam Medical Center, CHA University, Seoul
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No